CLINICAL TRIAL: NCT00772122
Title: Controlled Trial in Women With Recurrent Miscarriage of G-CSF Versus Placebo
Brief Title: Use of G-CSF for the Treatment of Unexplained Recurrent Miscarriage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Scarpellini Fabio, CERM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CERM0103
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Habitual Abortion
Keywords: Recurrent Miscarriage; G-CSF; pregnancy outcome; pregnancy outcome of pregnancies treated with G-CSF; treatment of recurrent miscarriage
MeSH Terms: conditions — Abortion, Habitual | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Granulocyte colony stimulating factor (Experimental): The G-CSF group of 35 women, underwent a daily sub-cutaneous administration of the filgrastim (Neupogen, Dompe', Italy), the recombinant G-CSF, at a dosage of 1 micro gram (100000 IU)/kg/day from the 6th day after ovulation till the occurrence of menstruation or to the end of the 9th week of gestation.
  Interventions: Drug: G-CSF
- placebo (saline solution) (Placebo Comparator): The placebo group consisting of 33 subjects, was given a treatment with saline solution at the 0.2ml/day subcutaneously/, from the 6th day after the ovulation till to the recurrence of menstrual loss or to the end of the 9th week.
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: G-CSF — daily sub-cutaneous administration of the recombinant G-CSF, at a dosage of 1 microgram (100000 IU)/kg/day from the 6th day after ovulation till the occurrence of menstruation or to the end of the 9th week of gestation.
  Other Names: filgrastim (Neupogen, Dompe', Italy),
  Arms: Granulocyte colony stimulating factor
Drug: saline solution — daily sub-cutaneous administration of saline solution 0.2ml from the 6th day after the ovulation till to the recurrence of menstrual loss or to the end of the 9th week.
  Arms: placebo (saline solution)

SUMMARY:
In order to investigate the effectiveness of G-CSF in preventing embryo demise, the investigators administered this cytokine to women with recurrent miscarriage in a randomized controlled study compared to women treated with placebo. Sixty eight women with unexplained primary recurrent miscarriage, all of them with at least four consecutive abortions and negative for all clinical investigations were selected for this study. Patients were randomly treated with G-CSF, starting on the 6th day after ovulation, or with placebo.

DETAILED DESCRIPTION:
The patients with unexplained primary (no previous successful pregnancy) recurrent miscarriage (RM) referred to the Hungaria Center for Endocrinology and Reproductive Medicine between January 2000 to January 2007 were considered eligible for the study. The patients had to fulfil the following inclusion criteria: woman's age less than 39 years, more than 4 previous abortions, failure of a previous treatment for RM (immunoglobulin infusion), and they had to be negative for the all the known causes of RM The study was reviewed and approved by the Institutional Review Board, and the clinical study was conducted according to Italian law and the Declaration of Helsinki for Medical Research involving Human Subjects. A sample size calculation showed that a total of 32 patient per group were needed in order to have a difference of 33% between the two groups a for p<0.005 and a beta>0.80 A total of 72 patients were considered eligible for the study, and 68 of them agreed to participate, signing an informed consent form. All the patients were informed about the eventual potential risks of this treatment for the mother and the foetus, other than the lack of information about the developmental toxicity of G-CSF. The patients were randomized by means of a computer generated randomization number sequence. All the patients were informed about the therapy and they gave their written informed consent. They were randomly assigned to the two arms of the study, one to G-CSF treatment and the other to placebo administration; the patients were blind to which treatment they were assigned to. The G-CSF group of 35 women, underwent a daily sub-cutaneous administration of the filgrastim (Neupogen, Dompe', Italy), the recombinant G-CSF, at a dosage of 1 microgram (100000 IU)/kg/day from the 6th day after ovulation till the occurrence of menstruation or to the end of the 9th week of gestation. The placebo group consisting of 33 subjects, was given a treatment with subcutaneous saline solution at the dosage of 0.2 ml daily, and also in this case, from the 6th day after the ovulation till to the recurrence of menstrual loss or to the end of the 9th week. Primary outcome was considered the pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* four or more previous consecutive abortion,
* failed previous treatment with intravenous immunoglobulins
* negative to all clinical investigation for recurrent miscarriage

Exclusion Criteria:

* in the last abortion a fetal karyotype showing chromosomal abnormality
* previous successful pregnancy

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2000-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome | During the treatment

SECONDARY OUTCOMES:
Pregnancy complication, undesired effects | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Scarpellini, MD, Principal Investigator — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (1):
- CERM, Rome, Italy

REFERENCES:
- [Derived] Scarpellini F, Sbracia M. Use of granulocyte colony-stimulating factor for the treatment of unexplained recurrent miscarriage: a randomised controlled trial. Hum Reprod. 2009 Nov;24(11):2703-8. doi: 10.1093/humrep/dep240. Epub 2009 Jul 17. PMID 19617208